CLINICAL TRIAL: NCT05835115
Title: Development and Validation of a Deep Learning-based Myopia and Myopic Maculopathy Detection and Prediction System
Status: Completed | Type: Observational
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Beijing Friendship Hospital (Other); Peking Union Medical College Hospital (Other); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); First Affiliated Hospital of Kunming Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: 2022SQ023
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Myopia; Myopic Macular Degeneration
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The training dataset: The training dataset was comprised of data from a school-based, prospective cohort (the Shanghai Time Outside to Reduce Myopia [STORM] trial) and data from another population-based, prospective study, the High Myopia Registration Study (SCALE-HM), with annual follow-up. Participants of the two studies were divided into a training set (70%), a tuning set (10%), and an internal test set (20%), which were not duplicated by each other at the participant level.
  Interventions: Diagnostic Test: A deep learning-based myopia and myopic maculopathy detection and prediction system
- The internal validation dataset: The internal validation dataset was comprised of data from a school-based, prospective cohort (the Shanghai Time Outside to Reduce Myopia [STORM] trial) and data from another population-based, prospective study, the High Myopia Registration Study (SCALE-HM), with annual follow-up. Participants of the two studies were divided into a training set (70%), a tuning set (10%), and an internal test set (20%), which were not duplicated by each other at the participant level.
  Interventions: Diagnostic Test: A deep learning-based myopia and myopic maculopathy detection and prediction system
- The external validation dataset: To test the extrapolation capabilities of the deep learning sysyem, two independent datasets, the Joint Five-site Fundus Test (JFFT) and the Hong Kong Children Eye Study (HKCES), were applied as external test sets. The JFFT study, a multi-site dataset, contains cross-sectional data from Shanghai, Yunnan, Inner Mongolia, Xinjiang and Guangzhou. HKCES, a population-based cohort study of eye conditions in children aged 6-8 years.
  Interventions: Diagnostic Test: A deep learning-based myopia and myopic maculopathy detection and prediction system

INTERVENTIONS:
Diagnostic Test: A deep learning-based myopia and myopic maculopathy detection and prediction system — This deep learning system is capable of analyzing fundus images for myopia staging, myopic maculopathy detection, cycloplegic refraction estimation and prediction, and risk stratification of myopia and myopic maculopathy onset.

SUMMARY:
Myopia has become a global public health issue. Myopia affects the psychological health of children and adolescents and poses a financial burden. Therefore, early detection and prediction of children at a high risk of myopia development and progression are critical for precise and effective interventions. In this study, we developed a deep learning system DeepMyopia, based on fundus images with the following objectives: 1) to predict myopia onset and progression; 2) To detect myopic macular degeneration for AI-assisted diagnosis; 3) To predict the development of myopic macular degeneration; 4) evaluate its cost-effectiveness.

DETAILED DESCRIPTION:
Myopia has become a global public health issue. Myopia affects the psychological health of children and adolescents and poses a financial burden. Furthermore, as myopia progresses it increases the risk of ocular complications such as myopic macular degeneration, leading to irreversible visual impairment or even blindness. According to the World Health Organization , more than 1 billion people worldwide are living with vision impairment caused by myopia, hyperopia, and other problems due to late detection. Therefore, early detection and prediction of children at a high risk of myopia development and progression are critical for precise and effective interventions.

In this study, we developed a deep learning system DeepMyopia, based on fundus images with the following objectives: 1) to predict myopia onset and progression; 2) To detect myopic macular degeneration for AI-assisted diagnosis; 3) To predict the development of myopic macular degeneration; 4) evaluate its cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with fundus images in the Shanghai Child and Adolescent Large-scale Eye Study (SCALE) ;
2. Subjects with fundus images in the Shanghai Time Outside to Reduce Myopia [STORM] trial;
3. Subjects with fundus images in the High Myopia Registration Study [SCALE-HM]
4. Subjects with fundus images in the Shanghai Myopia Screening (SMS) Study;
5. Subjects with fundus images in the Beijing Children Eye Study
6. Subjects with fundus images in the First Affiliated Hospital of Kunming Medical University;
7. Subjects with fundus images at the Ophthalmology Department of the First Affiliated Hospital of Xinjiang Medical University;
8. Subjects with fundus images at the Ophthalmology Department of the Affiliated Hospital of Inner Mongolia Medical University;
9. Subjects with fundus images at Zhongshan Eye Centre, Sun Yat-sen University;
10. Subjects with fundus images in the Hong Kong Children Eye Study;

Exclusion Criteria:

* Participants with poor-quality fundus images

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The SCALE, a prospective, school-based study, includes all children aged 4 to 14 years in Shanghai.
  The SCALE-HM, a population-based, prospective, examiner-masked study, includes children and adolescents aged between 4 and 18 years with high myopia.
  The STORM trial, a school-based, prospective, examiner-masked, cluster-randomized trial, includes children aged 6 to 9 years.
  The SMS study is a school-based cross-sectional survey from Shanghai, including kindergarten and primary school students in Year 1 and 2.
  The Beijing Children Eye study included children who came to the outpatient clinic of Beijing Friendship Hospital.
  The JFFT study contains cross-sectional data from Shanghai, Yunnan, Inner Mongolia, Xinjiang and Guangzhou.
  The Hong Kong Children Eye Study is a population-based cohort study of eye conditions in children aged 6-8 years.
Sampling Method: Probability Sample
Enrollment: 30526 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
myopia staging detection possibility score | immediately after inputting the data
  output of myopia staging task
myopic maculopathy detection possibility score | immediately after inputting the data
  output of myopic maculopathy detection task
predicted spherical equivalent | immediately after inputting the data
  output of assessing spherical equivalent task
predicted future annual spherical equivalent | immediately after inputting the data
  output of predicting future spherical equivalent task
risk score of myopia and myopic maculopathy progression | immediately after inputting the data
  output of the progression of myopia and myopic maculopathy predicion task

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No